CLINICAL TRIAL: NCT04263051
Title: Evaluation of UCPVax Plus Nivolumab as Second Line Therapy in Advanced Non Small Cell Lung : a Randomized Non Comparative Phase II Trial
Brief Title: Evaluation of UCPVax Plus Nivolumab as Second Line Therapy in Advanced Non Small Cell Lung Cancer
Acronym: Optim-UCPVax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Bristol-Myers Squibb (Industry); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2019/451; CA209-7CM (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCPVax + Nivolumab (Experimental): UCPVax vaccine (0,5 mg)
  Nivolumab (480 mg)
  Interventions: Drug: UCPVax + Nivolumab
- Standard second line chemotherapy (Other): Standard second line chemotherapy at the choice of the investigator.
  This arm will permit to assess the good calibration of the hypothesis on the experimental arm.
  Interventions: Drug: standard chemotherapy

INTERVENTIONS:
Drug: UCPVax + Nivolumab — UCPVax will be administrated at day 1 of week 1 ; 2 ; 3 ; 5 ; 6 ; 7 and then week 13 and every 2 months until months 12.
  Nivolumab will be administrated at the dose of 480 mg at day 1 and then every 4 weeks until disease progression or unacceptable toxicity according to label.
  At the end of COMBO phase, nivolumab will be continued every 4 weeks for maximum 24 months from the first administration, until disease progression or unacceptable toxicity according to standard of care.
  Arms: UCPVax + Nivolumab
Drug: standard chemotherapy — Second line chemotherapy at the choice of the investigator
  Arms: Standard second line chemotherapy

SUMMARY:
Lung cancer is the most commonly diagnosed malignancy and the leading cause of cancer-related mortality both in men and women worldwide.

The past few years have demonstrated great progress in the field of tumor immunotherapy through agents that address mechanisms of immune escape notably, so called immune checkpoint inhibitors (ICB). Indeed, ICB have emerged as a fatal weapon in the anticancer treatment arsenal. Anti-PD-1 and anti-PD-L1 antibodies have shown promising results in several cancers including Non-small Cell Lung Cancer (NSCLC) patients. Although such ICB extend patient's survival compared with conventional systemic therapies, they fail to control cancer progression in a significant proportion of patients which can reach up to 50-60% in NSCLC. Recent literature highlights a range of factors involved in the heterogeneous responses and failures to ICB therapies. The challenge is how can ICB treatment efficacy be extended to majority patients? To respond to this question, to increase the success of immunotherapy, immuno-oncology community develops combinations approaches.

The aim of these project is to evaluate the efficacy of Nivolumab plus a novel CD4Th1 inducer anti-cancer vaccine in NSCLC patients.

Nivolumab (NIVO), which is an anti-PD-1 antibody, has shown promising results in 2nd line treatment for advanced NSCLC.

UCPVax is a therapeutic anti-cancer vaccine based on the telomerase-derived helper peptides designed to induce strong TH1 CD4 T cell responses in cancer patients (NCT02818426).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Histologically or cytologically confirmed advanced NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma, undifferentiated carcinoma or other)
* Advanced NSCLC cancer patient with progressive disease after a first line of combo chemotherapy plus anti-PD-1 or chemotherapy plus anti-PD-L1 combination
* Measurable disease defined according to iRECIST v1.1 guidelines
* Patients must have a mandatory treatment-free interval of at least 21 days following previous systemic anti-cancer treatments
* Patients who have received previous systemic anticancer treatment and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 with the exception of Grade 2 alopecia
* Performance status 0 or 1 on the ECOG scale
* Females must be using highly effective contraceptive measures and have a negative pregnancy test prior to the start of dosing if of childbearing potential, or must have evidence of non-childbearing potential. Females of childbearing potential should use reliable methods of contraception from the time of the screening until 5 months after discontinuing study treatment. Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 7 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 7 months after discontinuing study treatment.
* Registration in a national health care system.
* Ability to comply with the study protocol, in the Investigator's judgment

Exclusion Criteria:

* Diagnosis of additional malignancy within 2 years prior to the inclusion with the exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer
* Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment
* Patient under guardianship, curatorship or under the protection of justice
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, ascites or symptomatic fistula
* Known active central nervous system metastases and/or carcinomatous meningitis
* Uncontrolled brain metastases
* Presence of EGFR mutation, ALK or ROS1 translocation
* history of hyperprogression during first line treatment with chemotherapy plus immunotherapy
* Inadequate organ functions: known cardiac failure of unstable coronaropathy, respiratory failure, or uncontrolled infection or another life-risk condition
* Active or chronic hepatitis B or C and/or HIV positive or known history of active Covid-19 infection, or a known history of active Tuberculosis bacillus
* Any immunosuppressive therapy (i.e. corticosteroids >10mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy
* Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of Nivolumab formulation
* History of idiopathic or secondary pulmonary fibrosis or evidence of active pneumonitis requiring a systemic treatment with 28 days before the planned start of study therapy
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 4 weeks prior to initiation of study treatment
* Receipt of a live, attenuated vaccine within 4 weeks prior to the initiation of treatment or anticipation that such a live, attenuated vaccine will be required during the study
* Patients requiring oxygen therapy
* For patients with a known cardiac history or with cardiac events occurring after first-line chemoimmunotherapy: LEVF<40% ; troponin > ULN; BNP > ULN
* Inadequate hematology, hepatic, renal functions or others inadequate laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
6 months Progression-Free Survival (PFS) rate | 6 months after the date of initiation of treatment (1st day of 1st cycle of chemotherapy)
  PFS is defined by the duration from the date of initiation of the treatment to the disease progression (RECIST) or death from any cause whichever occurs first, censoring cases without progression at the date of last disease assessment.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU of Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Institut de Cancérologie Privé CCGM, Montpellier
  - CH Mulhouse, Mulhouse
  - CHU de Nîmes, Nîmes
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adotevi O, Dosset M, Galaine J, Beziaud L, Godet Y, Borg C. Targeting antitumor CD4 helper T cells with universal tumor-reactive helper peptides derived from telomerase for cancer vaccine. Hum Vaccin Immunother. 2013 May;9(5):1073-7. doi: 10.4161/hv.23587. Epub 2013 Jan 28. PMID 23357860
- [Background] Godet Y, Dosset M, Borg C, Adotevi O. Is preexisting antitumor CD4 T cell response indispensable for the chemotherapy induced immune regression of cancer? Oncoimmunology. 2012 Dec 1;1(9):1617-1619. doi: 10.4161/onci.21513. PMID 23264913